CLINICAL TRIAL: NCT04970524
Title: Aesthetic Evaluation of Free Gingival Graft Applied by Partial De-epithelialization and Free Gingival Graft Applied by Conventional Method: a Randomized Controlled Clinical Study
Brief Title: Comparison of Conventional Free Gingival Grafts With Partially De-epithelized Free Gingival Grafts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonca Naziker (Other)
Responsible Party: Sponsor-Investigator, Yonca Naziker, Principal investigator Yonca Naziker, Izmir Katip Celebi University
Organization: Izmir Katip Celebi University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020-TDU-DİŞF-0002
Record Dates: First submitted 2021-04-08; First posted 2021-07-21 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Gingival Recession
Keywords: Partial de-epithelialized free gingival graft
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group(conventional free gingival graft) (Experimental): Conventional free gingival grafts are applied to the areas of the patients determined by randomization as suggested by Sullivan and Atkins.
  Interventions: Procedure: Comparison of conventional free gingival graft versus partial free gingival graft
- test group(Partially de-epithelialized free gingival graft) (Experimental): Partial free gingival graft is applied to the areas of the patients determined by randomization. Unlike the control group, the epithelium on the graft was partially epithelialized.
  Interventions: Procedure: Comparison of conventional free gingival graft versus partial free gingival graft

INTERVENTIONS:
Procedure: Comparison of conventional free gingival graft versus partial free gingival graft — Conventional free gingival graft was applied to the area of the patient with attached gingival insufficiency determined by randomization.
  Clinical and aesthetic comparisons were made in the postoperative 1st, 3rd and 6th months.
  Arms: control group(conventional free gingival graft)
Procedure: Comparison of conventional free gingival graft versus partial free gingival graft — Partially de-epithelialized free gingival graft was applied to the other region of the patient with attached gingival insufficiency determined by randomization.
  Clinical and aesthetic comparisons were made in the postoperative 1st, 3rd and 6th months.
  Arms: test group(Partially de-epithelialized free gingival graft)

SUMMARY:
In this study, the conventional SDG method applied to increase the adherent gingival band and partial de-epithelialized SDG methods were evaluated in terms of aesthetics and color compatibility of the recipient area with adjacent tissues.

This study is a controlled double-blind clinical trial randomized by split-mouth, envelope method.Clinical parameters and aesthetic harmony were compared at postoperative 1st, 3rd and 6th months after surgical procedures.Color harmony evaluation was made in 2 different ways, both by photo analysis of a blind researcher using computer software and by visual evaluation of the same blind researcher.

DETAILED DESCRIPTION:
The primary aim of this split mouth randomized controlled clinical trial is to compare the partial de-epithelialized free gingival grafting technique with the conventional free gingival grafting technique from an aesthetic point of view. The secondary aim of the study is to evaluate both techniques in terms of periodontal clinical parameters.

This study is a controlled double-blind clinical trial randomized by split-mouth, envelope method. Fifteen patients with attached gingiva width ≤2 mm in the lower jaw bilateral canine and premolar regions were included in the study. De-epithelialized free gingival grafts were applied to the region determined by envelope randomization, and conventional free gingival grafts were applied to the other region. The areas of the patients with insufficient attached gingiva were photographed before the operation, post-op 1st, 3rd, and 6th months, and visual aesthetic evaluations were made with photo analyzes. Clinical parameters such as keratinized gingival width, probing pocket depth, and recession depths were recorded at baseline and at 6 months. Results were represented as mean ± standard deviation and median, and a p value of <0,05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Absence of known systemic disease
* Not using any medication that may affect the periodontal tissues or prolong the bleeding time
* Having not previously operated on the palate area, which is both the receiving area and the donor area.
* The depth of the probing sulcus of all teeth is <3 mm
* Whole mouth plaque index and gingival index scores <1
* The teeth in the operation area are vital
* Absence of caries and / or restoration on the root surfaces of the teeth in the operation area
* Lack of attached gingiva in opposite jaws

Exclusion Criteria:

* Pregnant or lactating women,
* Smoking individuals,
* Individuals under the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-05-05 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2021-02-04 (Actual)

PRIMARY OUTCOMES:
aesthetic evaluation of both surgical methods | change in post-op 6 months
  Aesthetic evaluation of both surgical methods was done by a blinded researcher by photo analysis. For photo analysis, photographs of the recipient area were taken at the beginning and 6 months after the operation with the help of Adobe Photoshop program and evaluated on these photographs.

SECONDARY OUTCOMES:
clinical parameters | change in post-op 6 months
  In the clinical evaluation of both surgical methods, keratinized tissue width parameters were calculated and compared at baseline and pot-op 6 months.

CONTACTS AND LOCATIONS:
Locations (1):
- İzmir Katip Çelebi University Faculty of dentistry, Periodontology department, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Naziker Y, Ertugrul AS. Aesthetic evaluation of free gingival graft applied by partial de-epithelialization and free gingival graft applied by conventional method: a randomized controlled clinical study. Clin Oral Investig. 2023 Jul;27(7):4029-4038. doi: 10.1007/s00784-023-05029-8. Epub 2023 Apr 28. PMID 37118334